CLINICAL TRIAL: NCT03114085
Title: Apatinib Combined With Capecitabine Compared With Apatinib in the Treatment of Advanced Non-resectable Hepatocellular Carcinoma
Brief Title: Apatinib Combined With Capecitabine Compared With Apatinib Treat Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Zeng Zhiming, Doctor, First Affiliated Hospital of Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRGX-001
Record Dates: First submitted 2017-03-31; First posted 2017-04-14 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Capecitabine; apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib Combined with Capecitabine (Experimental): Apatinib,500mg,once a day, orally (after breakfast),from day 1 to day 21 (including day 21) for continuous administration, every 21 days for one cycle. If after two dose adjustments, the subject still can not tolerate toxicity, he or she should be out of group; Capecitabine,1000mg/m2,twice a day (at intervals of 12 hours,equivalent to a total daily dose of 2000 mg / m2),orally,sustained 14 days, off for 7 days, every 21 days for a cycle. If after two dose adjustments, the subject still can not tolerate toxicity, he or she should be out of group.
  Interventions: Drug: Capecitabine; Drug: Apatinib
- Apatinib (Active Comparator): Apatinib,500mg,once a day, orally (after breakfast),from day 1 to day 21 (including day 21) for continuous administration, every 21 days for one cycle. If after two dose adjustments, the subject still can not tolerate toxicity, he or she should be out of group;
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1000mg/m2 po bid, d1-d14, every 21 days for a cycle;
  Other Names: Aibin
  Arms: Apatinib Combined with Capecitabine
Drug: Apatinib — Apatinib 500 mg po qd, d1-d21, every 21 days for one cycle
  Other Names: Aitan

SUMMARY:
It is an open,randomized,controlled study, and the purpose of this study is to observe and evaluate the efficacy and safety of Apatinib combined with Capecitabine in the treatment of patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study is the clinical study of Apatinib combined with Capecitabine compared with Apatinib in the treatment of advanced non-resectable Hepatocellular Carcinoma, the object is patients with advanced hepatocellular carcinoma,its purpose is to observe and evaluate the efficacy and safety of Apatinib Mesylate Tablets combined with Capecitabine in the treatment of patients with advanced hepatocellular carcinoma, its main primary endpoint is TTP (time to progression) while the secondary endpoint is OS (overall survival), ORR (objective response rate), DCR (disease control rate), serum alpha-fetoprotein (AFP) levels and quality of life. 170 patients will be enrolled and 1:1 randomized into two groups: Apatinib combined Capecitabine and Apatinib alone. Major safety indicators are Vital signs, laboratory indicators, adverse events (AE), serious adverse events (SAE), drug-related AE and SAE, and specific AE (such as hypertension, proteinuria, and hand-foot syndrome), according to NCI-CTCAE.

ELIGIBILITY:
.Inclusion Criteria:

* Age: ≥18-75 years old
* Recurrent / Metastatic non-resectable HCC patients who are in strict compliance with clinical diagnostic criteria of the Standard of Primary Liver Cancer Diagnosis and Treatment (2011 edition) or diagnosis by histopathology or cytology, and are unable to accept palliative surgery or radiotherapy, and have at least one measurable lesion (according to mRECIST, the measurable lesions spiral CT scan length ≥ 10mm or enlarged lymph node diameter ≥ 15mm); the largest tumor ≤ 10cm
* Child-Pugh liver function rating: A or better B (≤ 7 points)
* BCLC stage is B-C period
* ECOG PS score within 1 week before enrollment: 0-1 points
* Expected survival time ≥12 weeks
* The main organs function is normal, that is, meeting the following criteria:

Blood examination:

HB ≥ 90 g / L; ANC ≥ 1.5 × 109 / L; PLT ≥ 60 × 109 / L;

Biochemical examination:

ALB ≥ 29 g / L; ALT and AST < 2.5 ULN; TBIL ≤ 2ULN; Creatinine ≤ 1.5ULN; (Albumin and bilirubin two indicators can only have one for 2 points in Child-Pugh rating)

* Women of childbearing age shall undergo pregnancy tests within 7 days before enrollment
* People to be tested are volunteered to join the study and sign informed consent. They should have good compliance and are easy to follow-up

  .Exclusion Criteria:
* Patients with hepatic cholangiocarcinoma or mixed cell carcinoma or fibrous lamellar cell carcinoma; or at the same time with other untreated malignant tumors in the past (within 5 years), except for cured skin basal cell carcinoma and cervical carcinoma in situ
* Patients who are preparing for liver transplantation (except those who have undergone liver transplantation)
* Patients with high blood pressure, and it can't be reduced to normal range (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg) by antihypertensive drug therapy
* Patients with level two or above myocardial ischemia or myocardial infarction, or poor controlled arrhythmia (including QTc interval men ≥ 450 ms, female ≥ 470 ms)
* According to NYHA standard Ⅲ ~ Ⅳ grade cardiac insufficiency or cardiac color Doppler ultrasound examination: LVEF (left ventricular ejection fraction) <50%
* Have a variety of factors affecting oral drugs (such as can not swallow, chronic diarrhea and intestinal obstruction, significantly affect drug taking and absorption)
* There is a history of gastrointestinal bleeding or a clear tendency to gastrointestinal bleeding in the past 6 months, such as: esophageal varicose veins with bleeding risk, local active ulcer lesions. Fecal occult blood ≥ (++) can not be grouped, if fecal occult blood (+),endoscopy is required
* Abdominal fistula, gastrointestinal perforation or abdominal abscess appeared within 28 days of participating in the study
* Coagulation dysfunction (INR> 1.5 or prothrombin time (PT)> ULN + 4 seconds), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy
* Patients with central nervous system metastasis or brain metastases
* Patients who is suffering or had suffered pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severe impairment of lung function
* Urine test indicated urine protein ≥ ++ or confirmed 24 hours urine protein> 1.0 g
* A strong CYP3A4 inhibitor treatment was received within 7 days before the study, or a strong CYP3A4 inducer was received within 12 days before the study
* Pregnant or lactating women; fertility patients who are reluctant or unable to take effective contraceptive measures
* Patients with mental illness, or history of mental drug abuse
* Patients with bone metastases had received palliative radiotherapy (radiotherapy area> 5% bone marrow area) within 4 weeks before participating in the study
* Patients who are joint with HIV infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-05-20 (Estimated); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-05-20 (Estimated)

PRIMARY OUTCOMES:
time to progression | through study completion, an average of 2 years
  From the randomization to the time of tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Zeng, Master, Principal Investigator — Guangxi Medical University First Affiliated Hospital

IPD SHARING:
Plan to Share IPD: Undecided